CLINICAL TRIAL: NCT05956405
Title: Retraining of the Amygdala and Insula for the Treatment of Persistent Covid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Miguel Servet (Other)
Responsible Party: Principal Investigator, Javier Garcia Campayo, Principal Investigator, Hospital Miguel Servet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI23/315
Record Dates: First submitted 2023-07-20; First posted 2023-07-21 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Mental Health Wellness
MeSH Terms: interventions — Air; Mindfulness

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amygdala & Insula Retraining + Mindfulness (Experimental)
  Interventions: Behavioral: AIR + Mindfulness
- Relaxation condition (Active Comparator)
  Interventions: Behavioral: Relaxation condition

INTERVENTIONS:
Behavioral: AIR + Mindfulness — AIR + Mindfulness program consists of 8 sessions of 120 minutes/session (10-12 people) Written material and sound recordings will be offered as support elements. The estimated duration of the program is two months.
  Arms: Amygdala & Insula Retraining + Mindfulness
Behavioral: Relaxation condition — Relaxation program consists of 8 sessions of 120 minutes/session (10-12 people) Written material and sound recordings will be offered as support elements. The estimated duration of the program is two months.
  Arms: Relaxation condition

SUMMARY:
Prolonged COVID, also known as post-COVID or Sar-CoV-2 infection with post-acute sequelae, refers to a set of multi-organ symptoms that persist in patients who have suffered SARS-CoV-2 infection, even after of the acute phase of the disease. Approximately 10% of people experience this set of symptoms after their acute COVID has resolved. Such symptoms may include respiratory problems, myalgia, extreme fatigue, moodiness, cognitive impairment, and difficulty sleeping.

Psychological therapies, such as mindfulness, have already demonstrated their effectiveness in pathologies of this type, improving mental health and physical function, as well as reinforcing acceptance and reducing symptoms. Specifically, amygdala-insula training was originally designed for patients with chronic fatigue syndrome as a method of reducing chronic over-sensitization and heightened fear response of the amygdala, which may be behind some of the symptoms related to both with this pathology as with fibromyalgia.

A lot of research is currently being done on different types of treatments such as pharmaceutical, biological, dietary, homeopathic and rehabilitation for the treatment of persistent COVID; however, an effective treatment has not yet been found. Therefore, this study aims to evaluate the impact of a retraining intervention of the amygdala and insula for the improvement of the quality of life of patients with persistent COVID.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-30 years old.
* Grant informed consent.
* Diagnosis of persistent COVID by primary care physicians.

Exclusion Criteria:

* Age: <18 years old
* Serious medical or psychiatric illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Short Form de 36 items (SF-36) | Baseline
  In the AIR + Mindfulness program group
Short Form de 36 items (SF-36) | Post-treatment 8 weeks from baseline
  In the AIR + Mindfulness program group
Short Form de 36 items (SF-36) | Three-months follow-up
  In the AIR + Mindfulness program group
Short Form de 36 items (SF-36) | Baseline
  In the relaxation program group
Short Form de 36 items (SF-36) | Post-treatment 8 weeks from baseline
  In the relaxation program group
Short Form de 36 items (SF-36) | Three-months follow-up
  In the relaxation program group

SECONDARY OUTCOMES:
Sociodemographic data Gender, age, marital status, education, occupation, economical level | Baseline
  In the AIR + Mindfulness program group
Sociodemographic data Gender, age, marital status, education, occupation, economical level | Baseline
  In the relaxation program group
Spanish Chronic Pain Grading Scale | Baseline
  In the AIR + Mindfulness program group
Spanish Chronic Pain Grading Scale | Baseline
  In the relaxation program group
Spanish Chronic Pain Grading Scale | Post-treatment 8 weeks from baseline
  In the AIR + Mindfulness program group
Spanish Chronic Pain Grading Scale | Post-treatment 8 weeks from baseline
  In the relaxation program group
Spanish Chronic Pain Grading Scale | Three-months follow-up
  In the AIR + Mindfulness program group
Spanish Chronic Pain Grading Scale | Three-months follow-up
  In the relaxation program group
Pain Catastrophizing Scale (PCS) | Baseline
  In the AIR + Mindfulness program group
Pain Catastrophizing Scale (PCS) | Baseline
  In the relaxation program group
Pain Catastrophizing Scale (PCS) | Post-treatment 8 weeks from baseline
  In the AIR + Mindfulness program group
Pain Catastrophizing Scale (PCS) | Post-treatment 8 weeks from baseline
  In the relaxation program group
Pain Catastrophizing Scale (PCS) | Three-months follow-up
  In the AIR + Mindfulness program group
Pain Catastrophizing Scale (PCS) | Three-months follow-up
  In the relaxation program group
Modified Fatigue Impact Scale (MFIS) | Baseline
  In the AIR + Mindfulness program group
Modified Fatigue Impact Scale (MFIS) | Baseline
  In the relaxation program group
Modified Fatigue Impact Scale (MFIS) | Post-treatment 8 weeks from baseline
  In the AIR + Mindfulness program group
Modified Fatigue Impact Scale (MFIS) | Post-treatment 8 weeks from baseline
  In the relaxation program group
Modified Fatigue Impact Scale (MFIS) | Three-months follow-up
  In the AIR + Mindfulness program group
Modified Fatigue Impact Scale (MFIS) | Three-months follow-up
  In the relaxation program group
Insomnia Severity Index (ISI) | Baseline
  In the AIR + Mindfulness program group
Insomnia Severity Index (ISI) | Baseline
  In the relaxation program group
Insomnia Severity Index (ISI) | Post-treatment 8 weeks from baseline
  In the AIR + Mindfulness program group
Insomnia Severity Index (ISI) | Post-treatment 8 weeks from baseline
  In the relaxation program group
Insomnia Severity Index (ISI) | Three-months follow-up
  In the AIR + Mindfulness program group
Insomnia Severity Index (ISI) | Three-months follow-up
  In the relaxation program group
General Anxiety Disorder-7 (GAD-7) | Baseline
  In the AIR + Mindfulness program group
General Anxiety Disorder-7 (GAD-7) | Baseline
  In the relaxation program group
General Anxiety Disorder-7 (GAD-7) | Post-treatment 8 weeks from baseline
  In the AIR + Mindfulness program group
General Anxiety Disorder-7 (GAD-7) | Post-treatment 8 weeks from baseline
  In the relaxation program group
General Anxiety Disorder-7 (GAD-7) | Three-months follow-up
  In the AIR + Mindfulness program group
General Anxiety Disorder-7 (GAD-7) | Three-months follow-up
  In the relaxation program group
Patient Health Questionnaire (PHQ-9) | Baseline
  In the AIR + Mindfulness program group
Patient Health Questionnaire (PHQ-9) | Baseline
  In the relaxation program group
Patient Health Questionnaire (PHQ-9) | Post-treatment 8 weeks from baseline
  In the AIR + Mindfulness program group
Patient Health Questionnaire (PHQ-9) | Post-treatment 8 weeks from baseline
  In the relaxation program group
Patient Health Questionnaire (PHQ-9) | Three-months follow-up
  In the AIR + Mindfulness program group
Patient Health Questionnaire (PHQ-9) | Three-months follow-up
  In the relaxation program group
Memory failures of Everyday (MFE) | Baseline
  In the AIR + Mindfulness program group
Memory failures of Everyday (MFE) | Baseline
  In the relaxation program group
Memory failures of Everyday (MFE) | Post-treatment 8 weeks from baseline
  In the AIR + Mindfulness program group
Memory failures of Everyday (MFE) | Post-treatment 8 weeks from baseline
  In the relaxation program group
Memory failures of Everyday (MFE) | Three-months follow-up
  In the AIR + Mindfulness program group
Memory failures of Everyday (MFE) | Three-months follow-up
  In the relaxation program group
Five Facets of Mindfulness Questionnaire (FFMQ) | Baseline
  In the AIR + Mindfulness program group
Five Facets of Mindfulness Questionnaire (FFMQ) | Baseline
  In the relaxation program group
Five Facets of Mindfulness Questionnaire (FFMQ) | Post-treatment 8 weeks from baseline
  In the AIR + Mindfulness program group
Five Facets of Mindfulness Questionnaire (FFMQ) | Post-treatment 8 weeks from baseline
  In the relaxation program group
Five Facets of Mindfulness Questionnaire (FFMQ) | Three-months follow-up
  In the AIR + Mindfulness program group
Five Facets of Mindfulness Questionnaire (FFMQ) | Three-months follow-up
  In the relaxation program group
Emotional Regulation Questionnaire (ERQ) | Baseline
  In the AIR + Mindfulness program group
Emotional Regulation Questionnaire (ERQ) | Baseline
  In the relaxation program group
Emotional Regulation Questionnaire (ERQ) | Post-treatment 8 weeks from baseline
  In the AIR + Mindfulness program group
Emotional Regulation Questionnaire (ERQ) | Post-treatment 8 weeks from baseline
  In the relaxation program group
Emotional Regulation Questionnaire (ERQ) | Three-months follow-up
  In the AIR + Mindfulness program group
Emotional Regulation Questionnaire (ERQ) | Three-months follow-up
  In the relaxation program group
Acceptance and Action Questionnaire-II (AAQ-II) | Baseline
  In the AIR + Mindfulness program group
Acceptance and Action Questionnaire-II (AAQ-II) | Baseline
  In the relaxation program group
Acceptance and Action Questionnaire-II (AAQ-II) | Post-treatment 8 weeks from baseline
  In the AIR + Mindfulness program group
Acceptance and Action Questionnaire-II (AAQ-II) | Post-treatment 8 weeks from baseline
  In the relaxation program group
Acceptance and Action Questionnaire-II (AAQ-II) | Three-months follow-up
  In the AIR + Mindfulness program group
Acceptance and Action Questionnaire-II (AAQ-II) | In the relaxation program group
  In the AIR + Mindfulness program group

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry. Miguel Servet University Hospital, Zaragoza, Spain

REFERENCES:
- [Derived] Gasion V, Barcelo-Soler A, Beltran-Ruiz M, Hijar-Aguinaga R, Camarero-Grados L, Lopez-Del-Hoyo Y, Garcia-Campayo J, Montero-Marin J. Effectiveness of an amygdala and insula retraining program combined with mindfulness training to improve the quality of life in patients with long COVID: a randomized controlled trial protocol. BMC Complement Med Ther. 2023 Nov 9;23(1):403. doi: 10.1186/s12906-023-04240-0. PMID 37946190